CLINICAL TRIAL: NCT05723198
Title: A Phase 3, Double-Blind, Randomized, Placebo-Controlled Trial to Evaluate the Efficacy, Safety, and Pharmacokinetics (PK) of Baricitinib in Children From 6 Years to Less Than 18 Years of Age With Alopecia Areata
Brief Title: A Study of Baricitinib (LY3009104) in Children From 6 Years to Less Than 18 Years of Age With Alopecia Areata
Acronym: BRAVE-AA-PEDS
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16875; I4V-MC-JAIO (Other: Eli Lilly and Company); 2022-502700-78-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-02-03; First posted 2023-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Areata Alopecia; Alopecia; Hypotrichosis; Hair Diseases; Skin Diseases; Pathological Conditions, Anatomical
MeSH Terms: conditions — Alopecia; Hypotrichosis; Hair Diseases; Skin Diseases; Pathological Conditions, Anatomical | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Baricitinib High Dose (Experimental): Participants will receive baricitinib high dose orally.
  Interventions: Drug: Baricitinib
- Baricitinib Low Dose (Experimental): Participants will receive baricitinib low dose orally.
  Interventions: Drug: Baricitinib
- Placebo (Placebo Comparator): Participants will receive placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Baricitinib — Administered orally
  Other Names: LY3009104
  Arms: Baricitinib High Dose; Baricitinib Low Dose
Drug: Placebo — Administered orally
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine the efficacy and safety of baricitinib for the treatment of severe or very severe alopecia areata (hair loss) in children from 6 years to less than 18 years of age.

The study is divided into 4 periods, a 5-week Screening period, a 36-week Double-Blind Treatment Period, an approximately 2-year Long-term Extension Period, and a 4-week Post-treatment Follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment will be fully sequential by age group, with adolescents (12 to less than 18 years old) enrolling before children (6 to less than 12 years old).
* Have severe areata alopecia (AA) for at least 1 year
* Diagnosis for at least 1 year
* Current AA episode of at least 6 months' duration
* SALT score ≥50% at screening and baseline
* History of trial and failure with at least 1 available treatment (topical or other) for AA
* History of psychological counseling related to AA
* Current episode of severe AA of less than 8 years.

  * Note: Participants who have severe AA for ≥8 years may be enrolled if episodes of regrowth, spontaneous or under treatment, have been observed on the affected areas over the past 8 years.

Exclusion Criteria:

* Primarily "diffuse" type of AA (characterized by diffuse hair shedding).
* Are currently experiencing other forms of alopecia including, but not limited to trichotillomania, telogen effluvium, chemotherapy-induced hair loss, or any other concomitant conditions (for example, tinea capitis, psoriasis, lupus erythematosus, or secondary syphilis) that would interfere with evaluations of the effect of study medication on AA.
* Are largely or wholly incapacitated permitting little or no self-care, such as being bedridden
* Have uncontrolled arterial hypertension
* Have had major surgery within 8 weeks prior to screening or will require major surgery during the study
* Have a history or presence of cardiovascular, respiratory, hepatic, gastrointestinal, endocrine, hematological, neurological, or neuropsychiatric disorders or any other serious and/or unstable illness that, in the opinion of the investigator, could constitute an unacceptable risk when taking IP or interfere with the interpretation of data.
* Have a positive test for hepatitis B virus (HBV) infection
* Have hepatitis C virus (HCV) infection (positive for anti hepatitis C antibody with confirmed presence of HCV ribonucleic acid [RNA]).
* Have evidence of human immunodeficiency virus (HIV) infection and/or positive HIV antibodies.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 595 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Achieving an Absolute Severity of Alopecia Tool (SALT) ≤20 | Week 36

SECONDARY OUTCOMES:
Percent Change from Baseline in SALT Score | Baseline, Week 36
Percentage of Participants Achieving At Least 90% Improvement from Baseline (SALT90) | Week 36
Percentage of Participants Achieving an Absolute SALT ≤10 | Week 36
Percentage of Participants with Patient Reported Outcome (PRO) for Scalp Hair Assessment Score of 0 or 1 Among Participants 12 Years and Older with PRO for Scalp Hair Assessment Score ≥3 at Baseline | Week 36
Mean Change from Baseline in SALT Score | Baseline, Week 36
Percentage of Participants Achieving At Least 50% Improvement from Baseline (SALT50) | Week 36
Percentage of Participants Achieving At Least 75% Improvement from Baseline (SALT75) | Week 36
Percentage of Participants Achieving At Least 100% Improvement from Baseline (SALT100) | Week 36
Percentage of Participants Achieving Clinician-Reported Outcome (ClinRO) Measure for Eyebrow (EB) Hair Loss 0 or 1 Among Participants with CLinRO Measure for EB Hair Loss ≥2 at Baseline | Week 36
Percentage of Participants Achieving ClinRO Measure for Eyelash (EL) Hair Loss 0 or 1 Among Participants with CLinRO Measure for EL Hair Loss ≥2 at Baseline | Week 36
Percentage of Participants Achieving PRO Measure for EB 0 or 1 (Among Participants 12 Years or Older with PRO Measure for EB ≥2 at Baseline) | Week 36
Percentage of Participants Achieving PRO Measure for EL 0 or 1 (Among Participants 12 Years or Older with PRO Measure for EL ≥2 at Baseline) | Week 36
Mean Change from Baseline in Hospital Anxiety Depression Scale (HADS) | Week 36
  The HADS is a participant-rated instrument used to assess both anxiety and depression and is available in a pediatric self-report for participants ≥12 years old. This instrument consists of 14 item questionnaires, each item is rated on a 4-point scale. Scores for each domain (anxiety and depression) can range from 0 to 21, with higher scores indicating greater anxiety or depression.
Mean Change from Baseline in Patient-Reported Outcome Measurement Information System (PROMIS) Anxiety Score | Baseline, Week 36
  The PROMIS Anxiety Short Form (8 questions, 8a v2.0) is available in a pediatric self-report (ages 8 to <18 years) and for parents/caregivers serving as proxy reporters for their children (youth ages ≥5 years). Both pediatric self-report and proxy-report versions assess anxiety "in the past seven days". Response options range from 1 = Never; 2 = Rarely; 3 = Sometimes; 4 = Often; to 5 = Almost always. Total raw scores are converted to T-Scores with higher scores representing greater anxiety.
Mean Change from Baseline in PROMIS Depression Score | Baseline, Week 36
  The PROMIS Depression Short Form (8a v2.0 and 6a v2.0) is available in a pediatric self-report (ages 8 to <18 years) and for parents/caregivers serving as proxy reporters for their children (youth ages ≥5 years). Both pediatric self-report and proxy-report versions assess depression "in the past seven days." Response options range from 1 = Never; 2 = Rarely; 3 = Sometimes; 4 = Often; to 5 = Almost always. Total raw scores are converted to T-Scores with higher scores representing greater depression.
Mean Change from Baseline in PROMIS Peer Relationship Score | Baseline, Week 36
  The PROMIS Peer Relationships Short Form planned to be used in the study measures 2 aspects of social functioning, friendship quality and peer acceptance, and is available in a pediatric self-report (ages 8 to <18 years) and for parents/caregivers serving as proxy reporters for their children (youth ages 5 to <8 years).
Mean Change from Baseline in Family Dermatology Life Quality Index (FDLQI) | Baseline, Week 36
  The FDLQI is a 10-item validated questionnaire designed for adult (>16 years old) family members of participants. The questionnaire is completed by family members of the AA participants (for example, parents/caregivers) and measures the secondary impact of the participant's skin disease on family QoL. Response categories include "not at all/not relevant," "only a little," "quite a lot," and "very much," with corresponding scores of 0, 1, 2, and 3, respectively, with unanswered ("not relevant") responses scored as 0.
Pharmacokinetics (PK): Maximum Concentration (Cmax) | Baseline through Week 36
PK: Area Under the Concentration Curve (AUC) | Baseline through Week 36
Change of Immunoglobulin G (IgG) Titers | Pre-Vaccination to 4 Weeks and 12 Weeks Post-Vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (127):
- United States (44):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Investigate MD, Scottsdale, Arizona
  - California Dermatology & Clinical Research Institute, Encinitas, California
  - Dermatology Research Associates, Los Angeles, California
  - University of California, San Diego/Rady Children's Hospital, San Diego - Pediatric & Adolescent Dermatology, San Diego, California
  - The Permanente Medical Group, Inc., San Francisco, California
  - Southern California Dermatology, Inc., Santa Ana, California
  - Dermatology Physicians of Connecticut, Fairfield, Connecticut
  - Skin Care Research, Inc, Boca Raton, Florida
  - Florida Academic Centers Research and Education, LLC, Coral Gables, Florida
  - D&H Doral Research Center LLC, Doral, Florida
  - Skin Care Research, Inc, Hollywood, Florida
  - Solutions Through Advanced Research, Inc., Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Pediatric Skin Research, LLC, Miami, Florida
  - Skin Care Physicians of Georgia, Macon, Georgia
  - Northwestern University, Chicago, Illinois
  - Northshore University Healthsystem, Skokie, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - The South Bend Clinic Center for Research, South Bend, Indiana
  - DermAssociates PC., Rockville, Maryland
  - Michigan Center for Research Company, Clarkston, Michigan
  - University of Minnesota Medical School, Minneapolis, Minnesota
  - MediSearch Clinical Trials, Saint Joseph, Missouri
  - Advanced Skin Research Center, Omaha, Nebraska
  - Montefiore Medical Center, The Bronx, New York
  - Dermatology Specialists of Charlotte, Charlotte, North Carolina
  - OnSite Clinical Solutions, Charlotte, North Carolina
  - Bexley Dermatology Research, Bexley, Ohio
  - Cincinnati Childrens Hospital Medical Center, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Vital Prospects Clinical Research Institute, P.C., Tulsa, Oklahoma
  - Northwest Dermatology Institute, Portland, Oregon
  - The Pennsylvania Centre for Dermatology, LLC, Exton, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - International Clinical Research - Tennessee (IC Research), Murfreesboro, Tennessee
  - Dermatology Treatment and Research Center, Dallas, Texas
  - Pediatric Dermatology of North Texas, Grapevine, Texas
  - Texas Dermatology and Laser Specialists, San Antonio, Texas
  - Complete Dermatology, Sugar Land, Texas
  - University of Utah MidValley Dematology, Murray, Utah
  - Virginia Clinical Research, Norfolk, Virginia
  - University of Wisconsin-Madison, Madison, Wisconsin
- Argentina (8):
  - Psoriahue Medicina Interdisciplinaria, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Derma Internacional SA, Buenos Aires
  - Buenos Aires Skin, Ciudad Autonoma Buenos Aires
  - Instituto de Neumonología Y Dermatología, Ciudad Autonoma Buenos Aires
  - Hospital Universitario Austral, Pilar
  - Centro Medico Privado de Reumatologia, SAN M. de Tucuman
  - Hospital del Niño Jesus, San Miguel de Tucumán
- Australia (4):
  - Skin and Cancer Foundation Australia - Darlinghurst Clinic, Darlinghurst
  - Sinclair Dermatology, Melbourne
  - Institute for Skin, Health, and Immunity, Mitcham
  - Veracity Clinical Research Pty Ltd, Wooloongabba
- Canada (6):
  - Dermatology Research Institute, Calgary
  - Skin Health, Cobourg
  - Lynderm Research Inc., Markham
  - Dr. Chih-ho Hong Medical Inc., Surrey
  - Research Toronto, Toronto
  - Wiseman Dermatology Research Inc., Winnipeg
- France (6):
  - CHRU de Brest - Hôpital Morvan, Brest
  - AP-HM CHU Timone - Pharmacie Secteur Essais Cliniques, Marseille
  - Centre Hospitalier Universitaire de Nantes - L' Hopital l'hôtel-Dieu, Nantes
  - Centre Hospitalier Universitaire de Nice - Hôpital l'Archet, Nice
  - Centre de Sante Sabouraud, Paris
  - Hôpital Clocheville Chru-Tours Département Dermatologie, Tours
- Germany (8):
  - Fachklinik Bad Bentheim, Bad Bentheim
  - Charite - Universitaetsmedizin Berlin - Campus Charite Mitte (CCM), Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Klinikum der Johann Wolfgang Goethe-Universität Frankfurt, Frankfurt am Main
  - Kath. Kinderkrankenhaus Wilhelmstift, Hamburg
  - Dermatologische Gemeinschaftspraxis Dres. Quist, Mainz
  - Klinikum Rechts der Isar der TU München, München
  - University of Muenster, Dept. of Dermatology, Central Study Coordination for innovative Dermatology, Münster
- Hungary (3):
  - Debreceni Egyetem Orvos-es Egészsegtudomanyi Centrum, Debrecen
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Pecsi Tudomanyegyetem, Pécs
- Japan (8):
  - Hamamatsu University Hospital, Hamamatsu
  - Kurume University Hospital, Kurume
  - Kyorin University Hospital, Mitaka
  - Rifu Dermatology Allergy Clinic, Miyagi-gun
  - Niigata University Medical & Dental Hospital, Niigata
  - Osaka City University Hospital, Osaka
  - Tokyo Medical University Hospital, Shinjuku-ku
  - Yamaguchi University Hospital, Ube
- Poland (14):
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk
  - CareClinic, Katowice
  - Centrum Medyczne Angelius Provita, Katowice
  - Gabinet Dermatologiczny, Kielce
  - Specjalistyczny Gabinet Dermatologiczny s.c., Krakow
  - Dermoklinika Centrum Medyczne s.c. M. Kierstan J. Narbutt A. Lesiak, Lodz
  - Kliniczny Szpital Wojewodzki Nr 1 im. Fryderyka Chopina w Rzeszowie, Rzeszów
  - DERMEDIC Jacek Zdybski, Swietokrzyski
  - Provita Poliklinika Sp. z o.o., Warsaw
  - Royalderm Agnieszka Nawrocka, Warsaw
  - Centralny Szpital Kliniczny MSWiA, Warsaw
  - Centrum Medyczne Evimed, Warsaw
  - Klinika Ambroziak Sp. Z.O.O., Warsaw
  - CityClinic Przychodnia Lekarsko-Psychologiczna, Wroclaw
- South Korea (14):
  - Pusan National University Hospital, Busan
  - Dankook University Hospital, Cheonan-si
  - Chungnam national university hospital, Daejeon
  - Inha University Hospital, Incheon
  - Jeonbuk National University Hospital, Jeonju
  - Kyungpook National University Hospital, Junggu
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Konkuk University Medical Center, Seoul
  - Kyunghee University Hospital at Gangdong, Seoul
  - Chung-Ang University College of Medicine - Chung-Ang University Hospital (CAUH), Seoul
  - Ajou University Hospital, Suwon
- Spain (6):
  - Hospital Universitario Germans Trias i Pujol, Badalona
  - Parc de Salut Mar - Hospital del Mar, Barcelona
  - Hospital Universitario Basurto, Bilbao (Bizkaia)
  - Clinica Pedro Jaen, Madrid
  - Hospital Universitario Infanta Leonor-INTERNAL MED, Madrid
  - Hospital General Universitario de Valencia, Valencia
- Taiwan (6):
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - Chung Shan Medical University Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Baricitinib (LY3009104) in Children From 6 Years to Less Than 18 Years of Age With Alopecia Areata — https://trials.lilly.com/en-US/trial/387275